CLINICAL TRIAL: NCT05675449
Title: A PHASE 1B, OPEN-LABEL STUDY OF ELRANATAMAB IN COMBINATION WITH CARFILZOMIB PLUS DEXAMETHASONE AND ELRANATAMAB IN COMBINATION WITH PF-07901801 IN PARTICIPANTS WITH RELAPSED REFRACTORY MULTIPLE MYELOMA
Brief Title: A Clinical Trial of Four Medicines (Elranatamab Plus Carfilzomib and Dexamethasone or Maplirpacept) in People With Relapsed Refractory Multiple Myeloma
Acronym: MagnetisMM-20
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C1071020; MAGNETISMM-20 (Other: Alias Study Number)
Record Dates: First submitted 2022-12-07; First posted 2023-01-09 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: elranatamab; relapsed; RRMM; BCMA; C1071020; MagnetisMM; maplipacelt; PF-06863135; carfilzomib; Bispecific antibody; PF-07901801; TTI-622; SIRPα; CD47
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 Dose Escalation (Experimental): Non randomized Elranatamab plus Carfilzomib and Dexamethasone
  Interventions: Drug: Elranatamab; Drug: Carfilzomib
- Part 2A Dose Escalation (Experimental): Non randomized Elranatamab plus Maplirpacept
  Interventions: Drug: Elranatamab; Drug: Maplirpacept
- Part 2B Dose Randomization (Experimental): Randomized dose level Elranatamab plus Maplirpacept
  Interventions: Drug: Elranatamab; Drug: Maplirpacept

INTERVENTIONS:
Drug: Elranatamab — BCMA-CD3 bispecific antibody
  Other Names: PF-06863135
Drug: Carfilzomib — proteasome inhibitor
  Other Names: Kyprolis
  Arms: Part 1 Dose Escalation
Drug: Maplirpacept — CD47-SIRP alpha-directed
  Other Names: PF-07901801, TTI-622
  Arms: Part 2A Dose Escalation; Part 2B Dose Randomization

SUMMARY:
The main purpose of the study is to evaluate the safety and tolerability of the combination of elranatamab and carfilzomib and dexamethasone or elranatamab and maplirpacept.

There are 2 parts to this study. Part 1 will evaluate the safety and tolerability of elranatamab when given in combination with carfilzomib plus dexamethasone. Part 2 has 2 arms. The first will evaluate the safety and tolerability of elranatamab when given in combination with maplirpacept. The second will identify the optimal dose(s) of elranatamab plus maplirpacept.

All study medicines are given over 4-week cycles. Everyone taking part in this study will receive elranatamab as a shot under the skin. Participants in Part 1 will also receive weekly carfilzomib as an IV infusion (given directly into a vein) and dexamethasone either by mouth (as a pill) or by IV infusion. Participants in Part 2 will receive elranatamab in combination with maplirpacept as an IV infusion (given directly into a vein)

The investigators will examine the experiences of people receiving the study medicines. This will help determine if the study medicines are safe and can be used for multiple myeloma treatment. Participants will take part in this study for about 2 years after the first dose.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of multiple myeloma as defined by IMWG criteria.
* Measurable disease based on IMWG criteria as defined by at least 1 of the following:

  * Serum M-protein ≥0.5 g/dL.
  * Urinary M-protein excretion ≥200 mg/24 hours.
  * Serum immunoglobulin FLC ≥10 mg/dL (≥100 mg/L) AND abnormal serum immunoglobulin kappa to lambda FLC ratio (<0.26 or >1.65).
* Part 1: Received at least 1 but not more than 3 prior lines of therapy for multiple myeloma (induction therapy followed by stem cell transplant and consolidation/maintenance therapy will be considered as 1 line of therapy).
* Part 2: Received at least 3 prior lines of therapy for multiple myeloma who are refractory to at least one IMiD, one PI and one anti-CD38 antibody.
* ECOG performance status 0-1.
* Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade ≤1.
* Not pregnant or breastfeeding and willing to use contraception.

Exclusion Criteria:

* Plasma cell leukemia, Smouldering MM, Waldenströms macroglobulinemia, Amyloidosis, POEMS Syndrome, Primary refractory MM
* Impaired cardiovascular function or clinically significant cardiovascular diseases.
* Participants with any active, uncontrolled bacterial, fungal, or viral infection.
* Stem cell transplant within 12 weeks prior to enrollment, or active graft versus host disease.
* Any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ.
* Part 1: Previous treatment with a BCMA-directed therapy.
* Part 2: Previous treatment with any anti-BCMA directed therapy, with the exception of CAR-T. Previous treatment with a CD47-SIRP alpha-directed therapy.
* Part 1: Prior treatment with carfilzomib
* Live attenuated vaccine within 4 weeks of the first dose of study intervention.
* Administration with an investigational product (e.g. drug or vaccine) concurrent with study intervention or within 30 days preceding the first dose of study intervention used in this study.
* Any of the following within 3 months of enrollment: erosive esophagitis, treatment resistant peptic ulcer, infectious or inflammatory bowel disease, pulmonary embolism or uncontrolled thromboembolic event.
* Intolerance to or participants who have had a severe (Grade ≥3) allergic or anaphylactic reaction to antibodies or therapeutic proteins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2026-04-22 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Part 1 Number of participants with dose limiting toxicity (DLT) | From first dose of elranatamab through the end of the first cycle of combination treatment, about 42 days.
  Dose limiting toxicity rate based on dose limiting toxicity evaluable participants.
Part 2A Number of participants with dose limiting toxicity | From the first dose of maplirpacept through the first cycle of combination treatment, about 64 days.
  Dose limiting toxicity based on dose limiting toxicity evaluable participants.
Part 2B Number of participants with dose limiting Toxicity | From first dose of elranatamab through the first cycle of combination treatment, about 42 days.
  Dose limiting toxicity rate based on dose limiting toxicity evaluable participants.

SECONDARY OUTCOMES:
Part 1: Number of Participants with Treatment Emergent Adverse Events (TEAE) by Seriousness and Relationship to Treatment | Assessed from baseline up to 90 days after last dose of study treatment.
  Counts of participants who had TEAEs, defined as newly occurring or worsening after first dose. Relatedness to study drug was assessed by the investigator. Participants with multiple occurrences of an AE within a category were counted once within the category.
Part 1: Number of Participants with Adverse Events (AE) characterized by type, frequency, severity. | Assessed from baseline up to 90 days after last dose of study treatment.
  An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Part 1: Number of Participants with Clinically Significant Change From Baseline in Laboratory Abnormalities | Accessed from baseline up to 90 days after the last dose of study treatment.
  Laboratory abnormalities as characterized by type, frequency, severity.
Part 1: Percent of participants with Best Overall Response (BOR) | Assessed for approximately 2 years
  BOR is defined as the best response recorded from treatment start until disease progression/recurrence based on International Myeloma Working Group (IMWG) response criteria.
Part 1: Percentage of Participants with an Objective Response Rate (ORR) | Assessed from enrollment for approximately 2 years.
  ORR rate is defined as the percent of participants having a Best Overall Response (BOR) of confirmed Stringent Complete Response (sCR), Complete Response (CR), Very Good Partial Response (VGPR), or Partial Response (PR) according to IMWG.
Part 1: Percentage of participants with a complete response rate (CRR) | Assessed for approximately 2 years
  Complete Response/ stringent Complete Response (CR+sCR) rate per IMWG response criteria as determined by investigator.
Part 1: Time to Response (TTR) | Assessed for approximately 2 years.
  TTR is defined, for participants with an objective response per IMWG criteria, as the time from the date of first dose to the first documentation of objective response that is subsequently confirmed.
Part 1: Duration of Response (DOR) | Assessed for approximately 2 years.
  DOR is defined, for participants with an objective response per IMWG criteria, as the time from the first documentation of objective response that is subsequently confirmed, until the first documentation of confirmed progressive disease (PD) per IMWG criteria.
Part 1: Duration of Complete Response (DOCR) | Assessed for approximately 2 years.
  DOCR is defined, for participants with a Complete Response/stringent Complete Response (CR+sCR) per IMWG criteria, as the time from the first documentation of CR/sCR that is subsequently confirmed, until the first documentation of confirmed progressive disease (PD) per IMWG criteria.
Part 1: Time of Progression Free Survival (PFS) | Assessed from enrollment until Progressive Disease or death for approximately 2 years.
  Progression free survival (IMWG response criteria)
Part 1: Time of Overall Survival (OS) | Assessed for approximately 2 years
  OS is the duration of time from first dose of study treatment to death.
Part 1: Minimal Residual Disease (MRD) Negativity Rate | Assessed for approximately 2 years
  MRD negativity rate is the proportion of participants acheiving CR+sCR with negative MRD, per IMWG sequencing criteria, from the date of first dose until the first documentation of confirmed progressive disease (PD), death or start of new anticancer therapy.
Part 1: Concentrations of carfilzomib | Once approximately 7 weeks from enrollment.
  Pre-dose and post-dose concentrations of cafilzomib
Part 1: Concentrations of elranatamab | Assessed for approximately 2 years.
  Pre-dose and post-dose concentrations of elranatamab
Part 1: Percentage of participants with positive anti-drug antibodies (ADA) against elranatamab | Assessed for approximately 2 years.
  Percent of participants with positive ADA to elranatamab when given in combination with carfilzomib and dexamethasone
Part 2A: Number of Participants with Treatment Emergent Adverse Events (TEAE) by Seriousness and Relationship to Treatment | Assessed from baseline up to 90 days after last dose of study treatment.
  Counts of participants who had TEAEs, defined as newly occurring or worsening after first dose. Relatedness to study drug was assessed by the investigator. Participants with multiple occurrences of an AE within a category were counted once within the category.
Part 2A: Number of Participants with Adverse Events (AE) characterized by type, frequency, severity. | Assessed from baseline up to 90 days after last dose of study treatment.
  An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Part 2A: Number of Participants with Clinically Significant Change From Baseline in Laboratory Abnormalities | Accessed from baseline up to 90 days after the last dose of study treatment.
  Laboratory abnormalities as characterized by type, frequency, severity.
Part 2A: Percent of participants with Best Overall Response (BOR) | Assessed for approximately 2 years
  BOR is defined as the best response recorded from treatment start until disease progression/recurrence based on International Myeloma Working Group (IMWG) response criteria.
Part 2A: Percentage of Participants with an Objective Response Rate (ORR) | Assessed from enrollment for approximately 2 years.
  ORR rate is defined as the percent of participants having a Best Overall Response (BOR) of confirmed Stringent Complete Response (sCR), Complete Response (CR), Very Good Partial Response (VGPR), or Partial Response (PR) according to IMWG.
Part 2A: Percentage of participants with a complete response rate (CRR) | Assessed for approximately 2 years
  Complete Response/ stringent Complete Response (CR+sCR) rate per IMWG response criteria as determined by investigator.
Part 2A: Time to Response (TTR) | Assessed for approximately 2 years.
  TTR is defined, for participants with an objective response per IMWG criteria, as the time from the date of first dose to the first documentation of objective response that is subsequently confirmed.
Part 2A: Duration of Response (DOR) | Assessed for approximately 2 years.
  DOR is defined, for participants with an objective response per IMWG criteria, as the time from the first documentation of objective response that is subsequently confirmed, until the first documentation of confirmed progressive disease (PD) per IMWG criteria.
Part 2A: Duration of Complete Response (DOCR) | Assessed for approximately 2 years.
  DOCR is defined, for participants with a Complete Response/stringent Complete Response (CR+sCR) per IMWG criteria, as the time from the first documentation of CR/sCR that is subsequently confirmed, until the first documentation of confirmed progressive disease (PD) per IMWG criteria.
Part 2A: Time of Progression Free Survival (PFS) | Assessed from enrollment until Progressive Disease or death for approximately 2 years.
  Progression free survival (IMWG response criteria)
Part 2A: Time of Overall Survival (OS) | Assessed for approximately 2 years
  OS is the duration of time from first dose of study treatment to death.
Part 2A: Minimal Residual Disease (MRD) Negativity Rate | Assessed for approximately 2 years
  MRD negativity rate is the proportion of participants achieving CR+sCR with negative MRD, per IMWG sequencing criteria, from the date of first dose until the first documentation of confirmed progressive disease (PD), death or start of new anticancer therapy.
Part 2A: Concentrations of maplirpacept | Assessed for approximately 2 years.
  Pre-dose and post-dose concentrations of maplirpacept
Part 2A: Concentrations of elranatamab | Assessed for approximately 2 years.
  Pre-dose and post-dose concentrations of elranatamab
Part 2A: Percentage of participants with positive anti-drug antibodies (ADA) against elranatamab | Assessed for approximately 2 years.
  Percent of participants with positive ADA to elranatamab when given in combination with maplirpacept
Part 2A: Percentage of participants with positive anti-drug antibodies (ADA) against maplirpacept | Assessed for approximately 2 years.
  Percent of participants with positive ADA to elranatamab when given in combination with elranatamab
Part 2B: Number of Participants with Treatment Emergent Adverse Events (TEAE) by Seriousness and Relationship to Treatment | Assessed from baseline up to 90 days after last dose of study treatment.
  Counts of participants who had TEAEs, defined as newly occurring or worsening after first dose. Relatedness to study drug was assessed by the investigator. Participants with multiple occurrences of an AE within a category were counted once within the category.
Part 2B: Number of Participants with Adverse Events (AE) characterized by type, frequency, severity. | Assessed from baseline up to 90 days after last dose of study treatment.
  An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Part 2B: Number of Participants with Clinically Significant Change From Baseline in Laboratory Abnormalities | Accessed from baseline up to 90 days after the last dose of study treatment.
  Laboratory abnormalities as characterized by type, frequency, severity.
Part 2B: Percent of participants with Best Overall Response (BOR) | Assessed for approximately 2 years
  BOR is defined as the best response recorded from treatment start until disease progression/recurrence based on International Myeloma Working Group (IMWG) response criteria.
Part 2B: Percentage of Participants with an Objective Response Rate (ORR) | Assessed from enrollment for approximately 2 years.
  ORR rate is defined as the percent of participants having a Best Overall Response (BOR) of confirmed Stringent Complete Response (sCR), Complete Response (CR), Very Good Partial Response (VGPR), or Partial Response (PR) according to IMWG.
Part 2B: Percentage of participants with a complete response rate (CRR) | Assessed for approximately 2 years
  Complete Response/ stringent Complete Response (CR+sCR) rate per IMWG response criteria as determined by investigator.
Part 2B: Time to Response (TTR) | Assessed for approximately 2 years.
  TTR is defined, for participants with an objective response per IMWG criteria, as the time from the date of first dose to the first documentation of objective response that is subsequently confirmed.
Part 2B: Duration of Response (DOR) | Assessed for approximately 2 years.
  DOR is defined, for participants with an objective response per IMWG criteria, as the time from the first documentation of objective response that is subsequently confirmed, until the first documentation of confirmed progressive disease (PD) per IMWG criteria.
Part 2B: Duration of Complete Response (DOCR) | Assessed for approximately 2 years.
  DOCR is defined, for participants with a Complete Response/stringent Complete Response (CR+sCR) per IMWG criteria, as the time from the first documentation of CR/sCR that is subsequently confirmed, until the first documentation of confirmed progressive disease (PD) per IMWG criteria.
Part 2B: Time of Progression Free Survival (PFS) | Assessed from enrollment until Progressive Disease or death for approximately 2 years.
  Progression free survival (IMWG response criteria)
Part 2B: Time of Overall Survival (OS) | Assessed for approximately 2 years
  OS is the duration of time from first dose of study treatment to death.
Part 2B: Minimal Residual Disease (MRD) Negativity Rate | Assessed for approximately 2 years
  MRD negativity rate is the proportion of participants achieving CR+sCR with negative MRD, per IMWG sequencing criteria, from the date of first dose until the first documentation of confirmed progressive disease (PD), death or start of new anticancer therapy.
Part 2B: Concentrations of maplirpacept | Assessed for approximately 2 years.
  Pre-dose and post-dose concentrations of maplirpacept
Part 2B: Concentrations of elranatamab | Assessed for approximately 2 years.
  Pre-dose and post-dose concentrations of elranatamab
Part 2B: Percentage of participants with positive anti-drug antibodies (ADA) against elranatamab | Assessed for approximately 2 years.
  Percent of participants with positive ADA to elranatamab when given in combination with maplirpacept
Part 2B: Percentage of participants with positive anti-drug antibodies (ADA) against maplirpacept | Assessed for approximately 2 years.
  Percent of participants with positive ADA to elranatamab when given in combination with elranatamab

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (39):
- United States (32):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Clinical Research Advisors (Encino Satellite Location), Encino, California
  - Clinical Research Advisors (Korea Town Satellite Location), Los Angeles, California
  - Clinical Research Advisors (West Hollywood Satellite Location), Los Angeles, California
  - Sylvester Comprehensive Cancer Center - Aventura, Aventura, Florida
  - Sylvester Comprehensive Cancer Center- The Lennar Foundation Medical Center, Coral Gables, Florida
  - Sylvester Comprehensive Cancer Center - Coral Springs, Coral Springs, Florida
  - University of Miami Hospital and Clinics - Deerfield Beach, Deerfield Beach, Florida
  - Sylvester Comprehensive Cancer Center - Hollywood, Hollywood, Florida
  - Griffin Cancer Research Building (GCRB), Miami, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Miami Hospital and Clinics, Miami, Florida
  - Sylvester Comprehensive Cancer Center - Kendall, Miami, Florida
  - Sylvester Comprehensive Cancer Center - Plantation, Plantation, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Administration Office, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - State University of Iowa, Division of Sponsored Programs, Iowa City, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Oncology Investigational Drug Service,Department of Pharmacy Services, Baltimore, Maryland
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Johns Hopkins University Cancer Immunology/GI Oncology, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber/Mass General Brigham Cancer Care, Inc, Boston, Massachusetts
  - MSK Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center - David H. Koch Center for Cancer Care (74th Street)., New York, New York
  - Memorial Hospital for Cancer and Allied Diseases, New York, New York
  - Memorial Sloan Kettering Cancer Center - Main Campus, New York, New York
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Israel (7):
  - Rambam Health Care Campus, Haifa
  - Division of Hematology Hadassah Medical Center - Ein Kerem, Jerusalem
  - The Research Fund of Hadassah Medical Organization (R.A.), Jerusalem
  - Hematology Division Davidoff Center, Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1071020